CLINICAL TRIAL: NCT00574457
Title: Improving Cardiovascular Risk Prediction Using Hand-Held Carotid Ultrasonography Study
Brief Title: Improving Cardiovascular Risk Prediction Using Hand Held Carotid Ultrasonography Study
Acronym: MERC-CIMT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 133JT68
Record Dates: First submitted 2007-12-12; First posted 2007-12-17 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Atherosclerosis; Stroke
Keywords: Atherosclerosis; Cardiovascular Risk Prevention; Carotid Ultrasound; Handheld ultrasound; Office Practice; Carotid Intima Media Thickness; Carotid Plaque
MeSH Terms: conditions — Atherosclerosis; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects that meet the inclusion criteria invited (Other)
  Interventions: Other: Carotid Ultrasound

INTERVENTIONS:
Other: Carotid Ultrasound — All subjects that meet the inclusion criteria at each certified site will be invited to participate and go through the same intervention (questionaire-scan-post scan questionaire and 1 month follow up questionaire)

SUMMARY:
1) Research questions:

1a. Can non-sonographer health care professionals in a community medical office practice setting be trained to detect and evaluate subclinical atherosclerosis?

1b. Can carotid ultrasound performed in community office practices improve physician use of evidence-based, risk-reducing interventions and patient motivation to adhere to therapeutic recommendations?

DETAILED DESCRIPTION:
Health care providers from five medical practices will complete a 2-day training program that teaches instrumentation, scanning, measurement, quality assurance, and interpretation. They also will learn about CV risk assessment, intervention, and how to use an ultrasound-based CV risk stratification and treatment algorithm. After certification, each site will recruit 70 patients from their practice (total N=350). Subjects will complete their routine office visit and a pre-test survey designed to assess motivation and intention to change. The physician's initial plan of action based on usual care will be recorded. Next, the subject will have a standardized CV risk carotid ultrasound. The physician will revise his/her treatment plan based on the scan results and an ultrasound-based risk assessment algorithm that includes CV risk factors and ultrasound data. Evidence-based treatment recommendations for lifestyle changes and risk factor targets will be provided. The physician's scan-based plan of action will be recorded. The subject will be informed of the results and repeat the survey. All images, interpretations, and recommendations will be reviewed by the UW AIRP.

ELIGIBILITY:
Inclusion Criteria:

* Informed written consent from the subject prior to testing.
* Age ≥40 years old with at least 1 of the following risk factors for coronary artery disease.
* cigarette smoking
* diabetes mellitus
* hypertension (systolic blood pressure ≥140 mm Hg or taking antihypertensive medication)
* hyperlipidemia (low-density lipoprotein cholesterol ≥130 mg/dl or high-density lipoprotein cholesterol less than 40 mg/dl)
* family history of CV disease in a male first-degree relative <55 or a female first-degree relative <65 years old

Exclusion Criteria:

* Age >70 years
* Use of cholesterol-lowering medications in the past year
* Known active liver disease (AST or ALT >2x upper limit of normal in home lab)
* Known active thyroid disease (TSH outside normal limits in home lab)
* Uncontrolled hypertension (blood pressure >180/100 mmHg)
* Chronic kidney disease (on dialysis or known creatinine >2.5 mg/dL)
* History of coronary artery disease (previous myocardial infarction, coronary revascularization procedure, angina pectoris with documented ischemia)
* History of cerebrovascular disease (previous stroke, transient ischemic attack, or carotid revascularization procedure)
* History of peripheral arterial disease (claudication with abnormal ankle-brachial indices or previous revascularization procedure)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2007-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To determine if non-sonographer health care professionals working in a community medical office practice setting can be trained to detect and evaluate subclinical atherosclerosis. | 2 years

SECONDARY OUTCOMES:
To determine if carotid ultrasound performed in community office practices can improve physician use of evidence-based, risk-reducing interventions and if it can improve patient motivation to adhere to therapeutic recommendations. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James H Stein, MD, Principal Investigator — University of Wisconsin Medical School and Public Heath
Locations (5):
- United States (5):
  - Internal Medicine and Pediatrics, S.C., Fort Atkinson, Wisconsin
  - Mercy Clinic East, Janesville, Wisconsin
  - ProHealth Care Medical Centers, Oconomowoc, Wisconsin
  - Turke Family Medicine S.C., Watertown, Wisconsin
  - Moreland Family Medicine Associates, S.C., Waukesha, Wisconsin